CLINICAL TRIAL: NCT06246344
Title: Efficacy and Safety of Adaptive Boost Radiotherapy to Primary Lesions and Positive Nodes in the Neoadjuvant Treatment of Locally Advanced Rectal Cancer: a Prospective, Randomized, Controlled, Phase III Trial
Brief Title: Adaptive Boost Radiotherapy to Primary Lesions and Positive Nodes in the Neoadjuvant Treatment of Locally Advanced Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Other Study IDs: SDZLEC2023-390-01
Record Dates: First submitted 2024-01-28; First posted 2024-02-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: neoadjuvant; rectal cancer; chemoradiotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collecting surgical pathology specimens, fecal samples, and blood from patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-ART + non-boost: Radiotherapy: The pelvic lymph node drainage area (CTV) is targeted with a dose of 45-50 Gy delivered in 25 fractions.
  Concurrent Chemotherapy: During radiotherapy, concurrent administration of capecitabine at a dose of 825 mg/m2, twice daily.
  Consolidation Chemotherapy Phase: On Day 1, two cycles of the CAPEOX regimen are administered (capecitabine 1.0 g/m2 po bid d1-14 + oxaliplatin 130 mg/m2, q3w). Initiated 7-10 days after completion of LCCRT.
  Surgical Phase: Commencing on Day 1, the patient undergoes Total Mesorectal Excision (TME) following consolidation chemotherapy.
  Interventions: Radiation: Long course non-ART radiotherapy; Drug: Concurrent chemotherapy; Drug: Consolidation Chemotherapy; Procedure: Total mesorectal excision (TME) surgery
- ART + Boost: ART Option 1 (SIB):
  GTVp+GTVn: A total dose of 60-65 Gy delivered in 25 fractions using a simultaneous integrated boost approach.
  CTV: A total dose of 45-50 Gy delivered in 25 fractions.
  ART Option 2 (SB):
  GTVp+GTVn: An initial hypofractionated boost with a total dose of either 9-12 Gy delivered in 3 fractions or 10 Gy delivered in 2 fractions.
  Concurrent Chemotherapy: During radiotherapy, concurrent administration of capecitabine at a dose of 825 mg/m2, twice daily.
  Consolidation Chemotherapy Phase: On Day 1, two cycles of the CAPEOX regimen are administered (capecitabine 1.0 g/m2 po bid d1-14 + oxaliplatin 130 mg/m2, q3w). Initiated 7-10 days after completion of LCCRT.
  Surgical Phase: Commencing on Day 1, the patient undergoes Total Mesorectal Excision (TME) following consolidation chemotherapy.
  Interventions: Radiation: Adaptive Boost Radiotherapy; Drug: Concurrent chemotherapy; Drug: Consolidation Chemotherapy; Procedure: Total mesorectal excision (TME) surgery

INTERVENTIONS:
Radiation: Adaptive Boost Radiotherapy — The choice of adaptive protocol and delivery system is based on individual tumor characteristics, patient anatomy and institutional capabilities. This approach provides flexibility in treatment planning while adhering to evidence-based dose constraints. Adaptive radiotherapy is delivered using one of the following advanced platforms: the Elekta Unity MRI Linac (MR-guided) or Varian Ethos (CBCT-guided), or the United Imaging uRT-linac 506c (FBCT-guided).
  ART Option 1 (simultaneous integrated boost, SIB):
  GTVp+GTVn: A total dose of 60-65 Gy delivered in 25 fractions using a simultaneous integrated boost approach.
  CTV: A total dose of 45-50 Gy delivered in 25 fractions.
  ART Option 2 (sequential boost, SB) GTVp+GTVn: An initial hypofractionated boost with a total dose of either 9-12 Gy delivered in 3 fractions or 10 Gy delivered in 2 fractions.
  CTV: Followed by standard fractionation delivering 45-50 Gy in 25 fractions.
  Other Names: ART-boost
  Groups: ART + Boost
Radiation: Long course non-ART radiotherapy — Conventional long-course radiotherapy administered in a non-adaptive manner without dose escalation. Treatment will be targeted to the pelvic lymphatic drainage region only. A total dose of 45-50 Gy will be delivered in 25 fractions over the course of treatment.
  Other Names: non-ART + non-boost
  Groups: Non-ART + non-boost
Drug: Concurrent chemotherapy — Capecitabine (825 mg/m2, po, twice daily)
Drug: Consolidation Chemotherapy — Following the completion of concurrent chemoradiotherapy, consolidation chemotherapy will commence 7 to 10 days later. Patients will receive two cycles of the CAPEOX regimen. Each cycle comprises: Capecitabine: 1.0 g/m² administered orally twice daily on days 1 through 14, and Oxaliplatin: 130 mg/m² administered intravenously on day 1.
Procedure: Total mesorectal excision (TME) surgery — Total mesorectal excision surgery

SUMMARY:
This is a multicenter, randomized, controlled phase III trial to evaluate the efficacy and safety of adaptive boost radiotherapy to the primary lesions and positive lymph nodes based on MR or CBCT or FBCT-guided adaptive radiotherapy in the neoadjuvant treatment of locally advanced rectal cancer.

DETAILED DESCRIPTION:
Locally advanced rectal cancer (LARC), typically stage II (cT3-4/N0) or stage III (cT1-4/N1-3), requires multimodal treatment. Surgical resection alone is associated with a high rate of local recurrence. Neoadjuvant chemoradiotherapy (nCRT) followed by total mesorectal excision (TME), on the other hand, can better control local recurrence in LARC patients. However, the overall pathological complete response (pCR) rate and clinical complete response (cCR) rate are still low, and there is an inconsistency between them, Therefore, the preservation of the anus is still a challenge. Optimizing neoadjuvant treatment strategies, including strategies such as increasing concurrent chemotherapy and increasing the dose of radiotherapy, is essential to improve tumor regression and anal preservation.

Radiotherapy is an important treatment for controlling local recurrence and downstaging LARC. A common cause of cancer recurrence in rectal cancer is that tumor cells metastasise nearby positive lymph nodes, such as the lateral pelvic lymph nodes These sites can serve as refuges where the cancer can regroup and either recur at the original site or spread to other areas. Various studies have also investigated the role of radiotherapy dose escalation in promoting tumor regression. Seldom have these studies examined dose escalation to both the primary lesions and positive lymph nodes. One of the major limiting factors is the tradeoff between destruction of the cancer itself and collateral damage to the neighboring healthy tissues. However, recent advances in the field have made great strides in overcoming this obstacle. Adaptive radiation therapy (ART), including magnetic resonance (MR)-guided, cone beam computed tomography (CBCT)-guided, and fan beam computed tomography (FBCT)-guided, allows direct imaging of the target and organs at risk (OAR), combined with optimization of the treatment plan for anatomical changes, to deliver high-quality dose escalation regimens to improve treatment response while protecting OAR such as the bladder, femoral heads, and small bowel.

We hypothesize that by implementing simultaneous integrated boost (SIB) or sequential boost (SB) radiotherapy to both the primary lesions and positive lymph nodes based on ART, we can improve the cCR and pCR rates without increasing surgical difficulty, while maintaining tolerable safety.

Against the above background, this study aims to conduct a multicenter, randomized, controlled phase III trial to evaluate the efficacy and safety of SIB or SB radiotherapy to the primary lesions and positive lymph nodes based on MR or CBCT or FBCT-guided ART in the neoadjuvant treatment of LARC. Eligible patients will be randomized 1:1 into experimental and control groups, both of which will undergo long course concurrent chemoradiotherapy (LCCRT), consolidation chemotherapy and TME surgery. During LCCRT, the experimental group will receive SIB or SB dose escalation based on MR or CBCT or FBCT-guided ART, while the control group will receive conventional dose without ART.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed rectal adenocarcinoma.
* Tumor located ≤10cm from the anal verge.
* Age ≥18 years.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1.
* Primary treatment-naive tumor confirmed by endorectal ultrasound (ERUS) or -
* Magnetic resonance imaging (MRI) as cT3-4/N+ according to the 8th edition of AJCC staging.
* Ability to provide tissue and blood samples for translational research.
* Anticipated survival of ≥6 months.
* Normal major organ function (within 14 days prior to enrollment) and suitability for receiving chemoradiotherapy.

Exclusion Criteria:

* History of prior chemotherapy, radiotherapy, or surgical treatment for rectal cancer, including transanal tumor resection.
* Locally recurrent rectal cancer.
* History of familial adenomatous polyposis.
* Active Crohn's disease or ulcerative colitis.
* Allergy or hypersensitivity history to 5-fluorouracil (fluorouracil) and/or oxaliplatin.
* History of difficulty or inability to take or absorb oral medications.
* Diagnosis of malignancy other than rectal cancer within the past 5 years (excluding completely cured basal cell carcinoma, squamous cell carcinoma of the skin, and/or in situ carcinoma treated with radical resection).
* Confirmed distant metastasis, i.e., cM1, through imaging or biopsy.
* History of pelvic radiotherapy.
* Pregnant or lactating women.
* Presence of any severe or uncontrollable systemic illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced rectal cancer
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
pCR | 1 year
  primary tumor achieved pathological complete response
surgical difficulty | 2 years
  The difficulty score of a surgery is calculated through a comprehensive assessment of the following indicators: surgical blood loss, surgical blood loss, pelvic fibrosis, pelvic fibrosis, degree of edema, number of anastomotic fistulas, and number of urinary dysfunctions.

SECONDARY OUTCOMES:
cCR | 2 years
  primary tumor achieved clinical complete response
3-year overal survival rate | 3 years
  The proportion of patients from the commencement of self-diagnosis to the time of death for any reason within 3 years
5-year overal survival rate | 5 years
  The proportion of patients from the commencement of self-diagnosis to the time of death for any reason within 5 years
3-year disease free suvival rate | 3 years
  The proportion of patients from the initiation of surgery to tumor recurrence or death within 3 years
5-year disease free suvival rate | 5 years
  The proportion of patients from the initiation of surgery to tumor recurrence or death within 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. Higher scores mean a worse outcome.
The Late Effects Normal Tissue/Subjective Objective Management Analytic (LENT/SOMA) system | 3 years
  The Late Effects Normal Tissue/Subjective Objective Management Analytic (LENT/SOMA) system for grading of side effects after radiotherapy was proposed, mainly including tenesmus, mucosal loss, sphincter control, stool frequency, pain, bleeding, ulceration, stricture, etc. Higher scores mean a worse outcome.
Quality of life assessment using the EORTC QLQ-C30 questionnaire | 3 year
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is a validated instrument designed to assess quality of life in cancer patients. It comprises 30 items divided into multi-item scales and single-item measures evaluating global health status/quality of life, various functioning domains (physical, role, emotional, cognitive, social), and a range of symptoms. Scores for each scale range from 0 to 100. For the global health status and functioning scales, higher scores indicate a better outcome, while for the symptom scales, higher scores indicate more severe symptoms and thus a worse outcome.
Quality of life assessment using the EORTC QLQ-CR29 questionnaire | 3 years
  The EORTC QLQ-CR29 is a validated colorectal cancer-specific quality of life instrument designed to complement the QLQ-C30 core questionnaire. It consists of 29 items assessing both functional aspects (e.g. body image and sexual functioning) and symptom domains specific to colorectal cancer. Scores for each domain are linearly transformed to a 0-100 scale. For the functional scales, higher scores indicate better quality of life, whereas for the symptom scales, higher scores indicate greater symptom burden and consequently worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Department of Radiation Oncology, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Gollins S, Sebag-Montefiore D. Neoadjuvant Treatment Strategies for Locally Advanced Rectal Cancer. Clin Oncol (R Coll Radiol). 2016 Feb;28(2):146-151. doi: 10.1016/j.clon.2015.11.003. Epub 2015 Nov 29. PMID 26645661
- [Background] van Gijn W, Marijnen CA, Nagtegaal ID, Kranenbarg EM, Putter H, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer: 12-year follow-up of the multicentre, randomised controlled TME trial. Lancet Oncol. 2011 Jun;12(6):575-82. doi: 10.1016/S1470-2045(11)70097-3. Epub 2011 May 17. PMID 21596621
- [Background] Lefevre JH, Mineur L, Kotti S, Rullier E, Rouanet P, de Chaisemartin C, Meunier B, Mehrdad J, Cotte E, Desrame J, Karoui M, Benoist S, Kirzin S, Berger A, Panis Y, Piessen G, Saudemont A, Prudhomme M, Peschaud F, Dubois A, Loriau J, Tuech JJ, Meurette G, Lupinacci R, Goasgen N, Parc Y, Simon T, Tiret E. Effect of Interval (7 or 11 weeks) Between Neoadjuvant Radiochemotherapy and Surgery on Complete Pathologic Response in Rectal Cancer: A Multicenter, Randomized, Controlled Trial (GRECCAR-6). J Clin Oncol. 2016 Nov 1;34(31):3773-3780. doi: 10.1200/JCO.2016.67.6049. PMID 27432930
- [Background] Fokas E, Schlenska-Lange A, Polat B, Klautke G, Grabenbauer GG, Fietkau R, Kuhnt T, Staib L, Brunner T, Grosu AL, Kirste S, Jacobasch L, Allgauer M, Flentje M, Germer CT, Grutzmann R, Hildebrandt G, Schwarzbach M, Bechstein WO, Sulberg H, Friede T, Gaedcke J, Ghadimi M, Hofheinz RD, Rodel C; German Rectal Cancer Study Group. Chemoradiotherapy Plus Induction or Consolidation Chemotherapy as Total Neoadjuvant Therapy for Patients With Locally Advanced Rectal Cancer: Long-term Results of the CAO/ARO/AIO-12 Randomized Clinical Trial. JAMA Oncol. 2022 Jan 1;8(1):e215445. doi: 10.1001/jamaoncol.2021.5445. Epub 2022 Jan 20. PMID 34792531
- [Background] Fernandez-Martos C, Garcia-Albeniz X, Pericay C, Maurel J, Aparicio J, Montagut C, Safont MJ, Salud A, Vera R, Massuti B, Escudero P, Alonso V, Bosch C, Martin M, Minsky BD. Chemoradiation, surgery and adjuvant chemotherapy versus induction chemotherapy followed by chemoradiation and surgery: long-term results of the Spanish GCR-3 phase II randomized trialdagger. Ann Oncol. 2015 Aug;26(8):1722-8. doi: 10.1093/annonc/mdv223. Epub 2015 May 8. PMID 25957330
- [Background] Camma C, Giunta M, Fiorica F, Pagliaro L, Craxi A, Cottone M. Preoperative radiotherapy for resectable rectal cancer: A meta-analysis. JAMA. 2000 Aug 23-30;284(8):1008-15. doi: 10.1001/jama.284.8.1008. PMID 10944647
- [Background] Ngan SY, Burmeister B, Fisher RJ, Solomon M, Goldstein D, Joseph D, Ackland SP, Schache D, McClure B, McLachlan SA, McKendrick J, Leong T, Hartopeanu C, Zalcberg J, Mackay J. Randomized trial of short-course radiotherapy versus long-course chemoradiation comparing rates of local recurrence in patients with T3 rectal cancer: Trans-Tasman Radiation Oncology Group trial 01.04. J Clin Oncol. 2012 Nov 1;30(31):3827-33. doi: 10.1200/JCO.2012.42.9597. Epub 2012 Sep 24. PMID 23008301
- [Background] Garcia-Aguilar J, Chow OS, Smith DD, Marcet JE, Cataldo PA, Varma MG, Kumar AS, Oommen S, Coutsoftides T, Hunt SR, Stamos MJ, Ternent CA, Herzig DO, Fichera A, Polite BN, Dietz DW, Patil S, Avila K; Timing of Rectal Cancer Response to Chemoradiation Consortium. Effect of adding mFOLFOX6 after neoadjuvant chemoradiation in locally advanced rectal cancer: a multicentre, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):957-66. doi: 10.1016/S1470-2045(15)00004-2. Epub 2015 Jul 14. PMID 26187751
- [Derived] Wang H, Zhang X, Leng B, Zhu K, Jiang S, Feng R, Dou X, Shi F, Xu L, Yue J. Efficacy and safety of MR-guided adaptive simultaneous integrated boost radiotherapy to primary lesions and positive lymph nodes in the neoadjuvant treatment of locally advanced rectal cancer: a randomized controlled phase III trial. Radiat Oncol. 2024 Sep 12;19(1):118. doi: 10.1186/s13014-024-02506-6. PMID 39267085